CLINICAL TRIAL: NCT06152952
Title: Evaluation of Rhomboid Flap Outcome in the Surgical Treatment of Recurrent Sacrococcygeal Pilonidal Sinus vs. Deep Suturing
Brief Title: Rhomboid Flap vs. Deep Suturing in Recurrent Pilonidal Sinus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Dify Kamal, Principal Investigator, Assiut University
Other Study IDs: pilonidal sinus
Record Dates: First submitted 2023-11-12; First posted 2023-12-01 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Pilonidal Sinus Infected
Keywords: Rhomboid flap; Deep suturing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 : The rhomboid flap Approach: The flap will be dissected deep to the gluteal fascia (subfascial level) so as to raise thick a fasciocutaneous flap. This will assure good vascularity of the flap without dead space. The rhomboid flap (CDEF) will be mobilized from the gluteal fascia and sutured without tension in three layers (gluteal fascia with 2/0 Vicryl, subcutaneous fat with 3/0 Vicryl, and the skin with 4/0 Prolene). As all sides will be equal in length, the flap fits in place without tension. A suction drain will be left behind and the wound will be dressed as usual. Pressure wound dressing will be applied and removed on the third postoperative day.
  Interventions: Procedure: The rhomboid flap approach
- Group 2 : The deep suturing approach: A vertical elliptical incision encompassing all pilonidal pits will be made and excision of the sinus will be carried out down to the level of the sacrococcygeal fascia. Tension will be released by a limited sharp dissection above the fascia. After haemostasis is ensured using electrocautery, a suction drain will be inserted through a separate incision, then the deep fascia will be approximated and the wound will be closed in layers using polyglactin 0 sutures. Finally, the skin will be closed with 2/0 polypropylene interrupted mattress sutures.
  Interventions: Procedure: The rhomboid flap approach

INTERVENTIONS:
Procedure: The rhomboid flap approach — The rhomboid flap Approach :
  The flap will be dissected deep to the gluteal fascia (subfascial level) so as to raise thick a fasciocutaneous flap. This will assure good vascularity of the flap without dead space. The rhomboid flap (CDEF) will be mobilized from the gluteal fascia and sutured without tension in three layers
  The deep suturing approach :
  A vertical elliptical incision encompassing all pilonidal pits will be made and excision of the sinus will be carried out down to the level of the sacrococcygeal fascia. T then the deep fascia will be approximated and the wound will be closed
  Other Names: The deep suturing approach

SUMMARY:
This prospective clinical trial aims to compare the perioperative outcomes of rhomboid flap versus deep suturing in the management of recurrent sacrococcygeal pilonidal disease.

DETAILED DESCRIPTION:
Pilonidal disease derives its name from Latin- pilus meaning "hair," and nidus meaning "nest" . The source of pilonidal disease is thought to be a deep intergluteal sulcus. It is widely accepted that the establishment of the pilonidal sinus results from the penetration of shed hair shafts through the skin, which ultimately leads to an acute or chronic infected site .

Pilonidal disease is largely considered a surgical disease, especially in acute instances with secondary infection and abscess. Infection or abscess requires incision and drainage. Definitive treatment is delayed the majority of the time if there is an acute infection or abscess until after the infection has been addressed. Surgical options for chronic disease are numerous and can include "pit picking," curettage, aspiration, unroofing, or surgical excision. Defects can be closed primarily, with flaps or grafts, or allowed to heal by secondary intention .

The most serious problem of the various surgical approaches proposed is the recurrence rate, ranging from 0% to 40% .

The surgical treatment of patients with recurrent disease does not differ from the surgical treatment of primary pilonidal disease. In case of a recurrence with an abscess, incision and drainage prevail, while in case of chronic recurrent disease, a flap based procedure may be indicated following sinus excision with scarring, like the rhomboid flap .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 18 and 60 years;
* Patients with one or two small inactive sinuses will be included for easier excisional procedures;
* Previous intervention for pilonidal disease whether surgical or non-surgical;

Exclusion Criteria:

1 - Patients with an acute abscess. 2- Patients with mall inactive pilonidal sinus disease. 3- Age beyond the previous limits. 4- Patients with primary pilonidal disease. 5- Refusal to participate in the study. 6- Unfit for anaesthesia and surgery. 7- Patients with malignant neoplasms or inflammatory bowel disease.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Diversity in population, some come from a rural environment and others from the city
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome of comparing the perioperative of rhomboid flap versus deep suturing in the management of recurrent sacrococcygeal pilonidal disease. | baseline
  Primary Outcome :
  Postoperative recurrence rate. Recurrence will be defined as the additional outbreak of signs and symptoms of pilonidal disease after a disease-free interval following complete wound healing

SECONDARY OUTCOMES:
Secondary Outcome (subsidiary)of comparing the perioperative of rhomboid flap versus deep suturing in the management of recurrent sacrococcygeal pilonidal disease. | baseline
  Secondary Outcome (subsidiary):
  1. Operative time.
  2. Postoperative pain.
  3. The incidence of other complications.
  4. Postoperative cosmetic outcome.
  5. The duration to walk, sit on toilet free from pain.
  6. The duration till complete daily activities.

OTHER OUTCOMES:
Data management and analysis (Details needed): | baseline
  Data collection Data will be collected by the principal investigator from Assiut University Hospital from.
  Computer software We will use SPSS version 26 for analyzing the data. Statistical tests Quantitative data will be presented as means ± SD. Categorical and binary variables will be tested using the χ 2 test and Fisher's exact test. Statistical significance will be assumed when p < 0.05.

REFERENCES:
- [Background] Esposito C, Cerulo M, Esposito G, Turco A, Borgogni R, Carulli R, Di Mento C, Del Conte F, Coppola V, Escolino M. Endoscopic Treatment of Pilonidal Sinus Disease in Children: A Systematic Review. J Laparoendosc Adv Surg Tech A. 2023 May;33(5):512-517. doi: 10.1089/lap.2022.0564. Epub 2023 Apr 6. PMID 37023403
- [Background] Konoplitskyi V, Shavliuk R, Dmytriiev D, Dmytriiev K, Kyrychenko O, Zaletskyi B, Olkhomiak O. Pilonidal disease: changes in understanding of etiology, pathogenesis and approach to treatment. Wiad Lek. 2019 Aug 31;72(8):1559-1565. PMID 32012508
- [Background] Harries RL, Alqallaf A, Torkington J, Harding KG. Management of sacrococcygeal pilonidal sinus disease. Int Wound J. 2019 Apr;16(2):370-378. doi: 10.1111/iwj.13042. Epub 2018 Nov 15. PMID 30440104
- [Background] Grabowski J, Oyetunji TA, Goldin AB, Baird R, Gosain A, Lal DR, Kawaguchi A, Downard C, Sola JE, Arthur LG, Shelton J, Diefenbach KA, Kelley-Quon LI, Williams RF, Ricca RL, Dasgupta R, St Peter SD, Somme S, Guner YS, Jancelewicz T. The management of pilonidal disease: A systematic review. J Pediatr Surg. 2019 Nov;54(11):2210-2221. doi: 10.1016/j.jpedsurg.2019.02.055. Epub 2019 Mar 19. PMID 30948198
- [Background] de Parades V, Bouchard D, Janier M, Berger A. Pilonidal sinus disease. J Visc Surg. 2013 Sep;150(4):237-47. doi: 10.1016/j.jviscsurg.2013.05.006. Epub 2013 Aug 1. PMID 23911903

DOCUMENTS (1):
  • Study Protocol (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT06152952/Prot_000.pdf